CLINICAL TRIAL: NCT00000121
Title: The Prism Adaptation Study (PAS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-20
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Esotropia
Keywords: strabismus
MeSH Terms: conditions — Esotropia; Strabismus | interventions — Eyeglasses

INTERVENTIONS:
Device: Prisms in Eyeglasses

SUMMARY:
To determine whether the preoperative use of prisms in eyeglasses can improve the outcome of surgery for acquired esotropia, a type of strabismus.

To determine whether patients who respond to prism adaptation by developing a new stable angle of -deviation have a better surgical result than do patients who do not respond to prism adaptation.

To determine whether patients who respond to prism adaptation are more accurately corrected by operating for the prism-adapted angle or the original angle of deviation.

To determine the usefulness of certain input variables (e.g., age at the time of surgery, size of the deviation, visual acuity, binocular function, refractive error) in predicting which patients are more likely to benefit from prism adaptation.

DETAILED DESCRIPTION:
Acquired esotropia (crossed eyes that develop after a child reaches the age of 6 months) accounts for 25 percent of all patients with misaligned eyes. Surgery to correct esotropia is done primarily to attain functional use of the two eyes together. The cosmetic aspect of the surgery is secondary. In 40 to 50 percent of cases, more than one operation is needed to accomplish the primary goal, and in some cases even three and four operations are needed.

Preliminary studies from two eye care centers reported that the use of prisms on eyeglasses for about a month before surgery led to good results after a single operation in more than 90 percent of patients. These uncontrolled preliminary studies pointed to the need for a multicenter, randomized, controlled clinical trial designed to prove or disprove scientifically the beneficial effect of prisms.

The Prism Adaptation Study was a double randomization trial involving 286 patients. Three-fifths of the patients were randomly selected for prism adaptation before surgery. Of the patients who responded to the prisms, one-half were randomly selected to have surgery based on the amount of prism required to stabilize the deviation, and the other half had surgery based on the amount of esotropia originally measured. Patients who did not respond to the prisms also had surgery based on the amount of esotropia measured, as did the two-fifths of the patients who did not undergo prism adaptation.

Patients were examined postoperatively at 1 week, 1 month, 3 months, 6 months, and 1 year. An independent examiner, masked to the treatment assignment, evaluated the patient at the 6-month followup. The results were analyzed to determine whether the outcome was better in patients who underwent prism adaptation or in those who underwent conventional treatment. Because the examiner did not know what type of treatment a patient had received, he or she would have no bias in evaluating the results.

ELIGIBILITY:
An eligible male or female must have been age 3 years or older (adults were included) and must have had esotropia that occurred at age 6 months or older, with no history of previous eye muscle surgery.

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 1984-03; Study Completion 1989-05 (Actual)

REFERENCES:
- [Background] Efficacy of prism adaptation in the surgical management of acquired esotropia. Prism Adaptation Study Research Group. Arch Ophthalmol. 1990 Sep;108(9):1248-56. doi: 10.1001/archopht.1990.01070110064026. PMID 2100986
- [Background] Repka MX, Connett JE, Scott WE. The one-year surgical outcome after prism adaptation for the management of acquired esotropia. Ophthalmology. 1996 Jun;103(6):922-8. doi: 10.1016/s0161-6420(96)30586-1. PMID 8643248